CLINICAL TRIAL: NCT01233427
Title: The Infant Feeding Experience of New Mothers - a Descriptive Pilot Study.
Brief Title: Infant Feeding Study.09-68
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 09-68
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Describe the Infant Feeding Attitudes; Intentions of a Sample of Expectant First-time Mothers; Estimate the Prevalence of Early Lactation Difficulties

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Characterize a population-based sample of first-time expectant mothers with regards to maternal metabolic health and their infant feeding experience.

DETAILED DESCRIPTION:
The long range purpose of this pilot study is to inform the development of an NIH-funded randomized intervention trial designed to improve early breastfeeding outcomes for mothers planning to breastfeed. The purpose of the pilot study is to 1) described the prenatal infant feeding attitudes and intentions of population-based sample of expectant mothers from the same recruitment base as the future intervention trial, 2) characterize the metabolic health profiles of the sample and 3) estimate the prevalence of early lactation difficulties among the subset of this sample that initiates breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* First-time expectant mother, speaks English, receiving OB care at designated practice group

Exclusion Criteria:

* 1) Under 18 years old; 2)no access to local telephone 3) multiple gestation 4) history of major breast surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: breastfeeding moms
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Early lactation difficulties | 1 year
  a)Estimate the prevalence of early lactation difficulties among the subset of this sample that initiates breastfeeding, b) examine the relationship between metabolic health and lactation difficulties

SECONDARY OUTCOMES:
Infant feeding attitudes | 1 year
  describe the prenatal infant feeding attitudes and intentions of a sample of expectant mothers from the same recruitment base as the future intervention trial

CONTACTS AND LOCATIONS:
Overall Officials: Laurie A Nommsen-Rivers, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati

REFERENCES:
- [Result] Nommsen-Rivers LA, Dolan LM, Huang B. Timing of stage II lactogenesis is predicted by antenatal metabolic health in a cohort of primiparas. Breastfeed Med. 2012 Feb;7(1):43-9. doi: 10.1089/bfm.2011.0007. Epub 2011 Apr 27. PMID 21524193